CLINICAL TRIAL: NCT04371692
Title: Prevalence of SARS-Cov2 Infection Among HCW in Lille University Hospital
Brief Title: Prevalence of COVID-19 Infection Among HCW in a French University Hospital
Acronym: EXPOCOVIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Fondation Santé Roquette (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020_35; 2020-A00951-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Sars-CoV2
Keywords: Prevalence; Health Care Workers; occupational exposure; environmental exposure; serological testing; RT-PCR
MeSH Terms: interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-risk: staff working in a unit specifically for patients infected or suspected of being infected with SARS-Cov2
  Interventions: Other: self-administered questionnaire; Diagnostic Test: SARS-Cov2 testing
- Medium- risk: staff working in a unit that can accommodate patients infected or suspected of being infected with SARS-Cov2, i.e., all care services that do not fall into the high-risk group.
  Interventions: Other: self-administered questionnaire; Diagnostic Test: SARS-Cov2 testing
- Low-risk: off-patient staff
  Interventions: Other: self-administered questionnaire; Diagnostic Test: SARS-Cov2 testing

INTERVENTIONS:
Other: self-administered questionnaire — Every weeks during 2 months, clinical and occupational questionnaire are performed among a cohort of HCW exposed to covid occupational exposure
  Other Names: a specifically designed self-administered questionnaire
Diagnostic Test: SARS-Cov2 testing — Every weeks during 2 month, SARS-Cov2 RT-PCR, serological testing are performed among a cohort of HCW exposed to covid occupational exposure

SUMMARY:
The objective of this study is to determine the prevalence of SARS-Cov2 infection among health care workers exposed of Lille University Hospital, to describe its evolution during the epidemic taking into account the influence of occupational and environmental exposure determinants.

ELIGIBILITY:
Inclusion Criteria:

- Health Care workers with or without symptoms suggestive of a COVID-19 infection

Exclusion Criteria:

* HCW working off-site at the CHU de Lille
* HCW on sick leave.
* HCW outside the Lille University Hospital temporarily coming as reinforcements in the context of the epidemic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care workers with or without symptoms suggestive of a COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
the prevalence of SARS- Cov2 infection Health Care Worker with or without symptoms suggestive of a COVID-19 infection | at 2 months

SECONDARY OUTCOMES:
the prevalence of SARS- Cov2 infection Health Care Worker with or without symptoms suggestive of a COVID-19 infection | once week during 2 months
Occupational exposures associated with the SARS-Cov2 infection | once week during 2 months
Environmental exposures associated with the SARS-Cov2 infection | once week during 2 months
immunologic status of health Care Worker | once week during 2 months
inflammatory biomarkers status of Health Care Worker | once week during 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Annie SOBASZEK, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France